CLINICAL TRIAL: NCT06653452
Title: Application of PET/MRI in the Evaluation of the Efficacy of Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-LARC-FAPI
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced Rectal Cancer (LARC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-FDG PET/CT and PET/MR, 68Ga-FAPI-04 PET/CT and PET/MR (Experimental): After patient enrollment, 68Ga-FAPI-04 PET/CT and PET/MR examinations are performed. Within 1 week before and after the examination, PET/CT and PET/MR is also performed in patients.
  Interventions: Diagnostic Test: 18F-FDG PET/CT and PET/MR scan, 68Ga-FAPI-04 PET/CT and PET/MR scan

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT and PET/MR scan, 68Ga-FAPI-04 PET/CT and PET/MR scan — Patients with Locally Advanced Rectal Cancer underwent 68Ga-FAPI-04 PET/CT and PET/MR scan after injection of 0.02 to 0.04 mCi/Kg×patient weight (Kg). Within 1 week before and after the examination, 18F-FDG PET/CT and PET/MR is completed.

SUMMARY:
This study plans to include LARC patients receiving neoadjuvant therapy at this center, conducting PET/CT and PET/MR examinations before treatment, and PET/MR examinations before surgery after neoadjuvant therapy. The changes in the lesion before and after treatment will be compared to evaluate the efficacy of neoadjuvant therapy, including: the relief situation of the rectal primary lesion ; lymph node metastasis; local infiltration around the tumor; peritoneal and other distant metastases , etc. The pathological relief diagnosed by surgical pathology is the gold standard, and the predictive efficacy of PET/MR will be evaluated, comparing the advantages and disadvantages of 18F-FDG and 68Ga-FAPI PET/MR, and comparing with traditional PET/CT and rectal MRI to explore the value of PET/MRI in predicting the efficacy of neoadjuvant therapy in LARC patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-75 years old; (2) ECOG score 0-2; (3) Pathologically confirmed as rectal adenocarcinoma; (4) The lower edge of the tumor is within 12cm from the anal edge; (5) Clinically staged as cT3-4N0M0 or cTanyN+M0; (6) Untreated patients who have not received radiotherapy, chemotherapy, and surgery, etc.; (7) Good liver and kidney function, can tolerate radiotherapy and surgery; (8) Patients and their families can understand the research plan, voluntarily participate in this research and sign the informed consent form.

Exclusion Criteria:

* (1) ECOG score > 2; (2) Patients with multiple primary colorectal cancers; (3) Patients with a history of other malignant tumors within the past 5 years (except for cured basal cell carcinoma, cervical carcinoma in situ, surgically treated localized prostate cancer, or surgically removed breast ductal carcinoma in situ); (4) Patients with intestinal obstruction, intestinal perforation, gastrointestinal bleeding, and other emergencies requiring emergency surgery; (5) Pregnant or lactating women; (6) Patients with a history of severe mental illness, immune diseases, and hormone medication; (7) Patients with contraindications for MRI, PET examination, radiotherapy, immunotherapy, or surgical treatment; (8) Patients who have participated in other clinical studies within the last 3 months; (9) Any other conditions deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance including sensitivity, specificity, accuracy | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
TNM stage changed by 68Ga-FAPI-04 PET/CT and PET/MR compared to 18F-FDG PET/CT and PET/MR. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China